CLINICAL TRIAL: NCT02696655
Title: Development and Feasibility Testing of a Behavioural Intervention Targeting Multiple Lifestyle Behaviours to Improve Long Term Outcomes Following Liver Transplantation
Brief Title: Lifestyle Intervention For Liver Transplantation
Acronym: LIFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 7526
Record Dates: First submitted 2015-10-12; First posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Liver Disease
Keywords: transplantation
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- liver transplant patients (Experimental): Patients will use a behavioural intervention to assess its usability
  Interventions: Behavioral: Behavioural intervention

INTERVENTIONS:
Behavioral: Behavioural intervention — Behavioural intervention administered by healthcare professionals targetting multiple lifestyle behaviours

SUMMARY:
(i) To develop a behavioural intervention that supports healthcare professionals to effectively deliver lifestyle behaviour change of patients undergoing liver transplantation

(ii) To assess the acceptability and feasibility of the behavioural intervention during routine practice

DETAILED DESCRIPTION:
BACKGROUND

Liver transplantation is the most effective treatment for decompensated chronic liver disease and is associated with improvements in life expectancy and quality of life(1). Recent advances in immunosuppressive therapy; greater surgical and anaesthetic expertise and optimised risk assessment procedures have shown to be associated with improvements in 90 day, 1 and 5 year survival (2). However, non-liver causes of death are on the increase with malignancy (22%), cardiovascular disease (11%), infection (9%) and renal failure (6%) becoming leading causes of death at one year (3)

It is well recognised that liver transplantation is associated with the onset of a number of conditions that increase risk of early mortality, including new onset diabetes, hypertension and dyslipidaemia (4,5). These conditions have the potential to be prevented or improved by behavioural intervention targeting health and lifestyle behaviours including physical activity, diet, smoking and medication adherence (6). Lifestyle factors are central to both survival on the waiting list and long-term post transplant survival. Therefore it is important to support patients to make positive and sustainable lifestyle behaviour changes. However, this represents a complex medical challenge because rarely are clinical teams trained to target lifestyle behaviour change in a meaningful/personalised way.

AIMS OF THE STUDY

The aim is to develop a behavioural intervention that can be used by all medical personnel involved in the care of patients being assessed for transplantation, whilst listed for transplantation and post transplantation to improve long-term outcomes. The intervention will be co-developed by clinicians and patients to ensure it is fit for purpose. Healthcare professionals will be trained to target a range of health and lifestyle behaviours using evidence-based behavioural strategies. It is hoped this will lead to improvements in long-term survival by reducing modifiable risk factors for mortality.

OBJECTIVES

This study will develop and assess acceptability and feasibility of a multifaceted behaviour change intervention. The intervention will be designed to train healthcare professionals to use behavioural strategies to target key lifestyle behaviours in the context of liver transplantation, and to equip patients with behavioural skills to make positive changes to a range of lifestyle behaviours. In reality, this could be the most cost effective model to be able to enable lifestyle change for transplant patients. These healthcare professionals are front line staff and work with high volumes of transplant patients.

PRIMARY RESEARCH QUESTION Is a multifaceted behavioural intervention co-developed by healthcare professionals and patients acceptable and feasible and can it be delivered faithfully during routine clinical practice?

Objectives The objectives of this study are:- i) To co-develop an evidence-based, multifaceted behavioural intervention for delivery during routine clinical consultations ii) To develop a training programme that equips clinicians with the knowledge, skills and confidence to deliver a behavioural intervention during routine clinical practice iii) To determine whether the behavioural intervention is acceptable and feasible to both healthcare professionals and patients iv) To assess whether the behavioural intervention can be delivered faithfully during routine clinical practice v) To optimise the behavioural intervention based on feedback from clinicians and patients.

vi) To assess whether the intervention impacts positively on clinical outcomes (e.g., blood pressure, HbA1c levels) vii) To inform the design of a large randomised controlled trial if appropriate

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Undergoing or planned to undergo liver transplant assessment, listed for liver transplantation or have undergone liver transplantation at the Freeman Hospital
* Willing to participate in the study and able to provide written informed consent

Exclusion Criteria:

* Patients who can't speak English and require the use of an interpreter.
* Those who do not attend the Freeman Hospital for follow up care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-11 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility testing of the intervention | 1 year
  Qualitative assessment of the behavioural intervention by focus groups and interviews with patients and healthcare professionals

SECONDARY OUTCOMES:
Exercise capacity | 1 year
  Assessed by pedometers (average steps per day taken assessed over one week)
Hypertension | 1 year
  Change in blood pressure from baseline
Weight | 1 year
  change in weight since baseline
Diabetes | 1 year
  change in HBA1c from baseline
renal dysfunction | 1 year
  change in estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Leah Avery, Principal Investigator — Newcastle University
Locations (1):
- Dept of perioperative and critical care medicine, Freeman Hospital, Newcastle upon Tyne, Tyne and Wear, United Kingdom

REFERENCES:
- [Result] Tsochatzis EA, Bosch J, Burroughs AK. Liver cirrhosis. Lancet. 2014 May 17;383(9930):1749-61. doi: 10.1016/S0140-6736(14)60121-5. Epub 2014 Jan 28. PMID 24480518
- [Result] Germani G, Theocharidou E, Adam R, Karam V, Wendon J, O'Grady J, Burra P, Senzolo M, Mirza D, Castaing D, Klempnauer J, Pollard S, Paul A, Belghiti J, Tsochatzis E, Burroughs AK. Liver transplantation for acute liver failure in Europe: outcomes over 20 years from the ELTR database. J Hepatol. 2012 Aug;57(2):288-96. doi: 10.1016/j.jhep.2012.03.017. Epub 2012 Apr 18. PMID 22521347
- [Result] Pfitzmann R, Nussler NC, Hippler-Benscheidt M, Neuhaus R, Neuhaus P. Long-term results after liver transplantation. Transpl Int. 2008 Mar;21(3):234-46. doi: 10.1111/j.1432-2277.2007.00596.x. Epub 2007 Nov 21. PMID 18031464
- [Result] Benhamou PY, Penfornis A. Natural history, prognosis, and management of transplantation-induced diabetes mellitus. Diabetes Metab. 2002 Jun;28(3):166-75. PMID 12149596
- [Result] Gisbert C, Prieto M, Berenguer M, Breto M, Carrasco D, de Juan M, Mir J, Berenguer J. Hyperlipidemia in liver transplant recipients: prevalence and risk factors. Liver Transpl Surg. 1997 Jul;3(4):416-22. doi: 10.1002/lt.500030409. PMID 9346772
- [Result] Luca L, Westbrook R, Tsochatzis EA. Metabolic and cardiovascular complications in the liver transplant recipient. Ann Gastroenterol. 2015 Apr-Jun;28(2):183-192. PMID 25830307